CLINICAL TRIAL: NCT07362459
Title: A Phase III, Randomized, Double-blind, Multicenter Clinical Study to Evaluate the Efficacy and Safety of SCTB14 Versus Pembrolizumab as First-Line Therapy in Patients With Driver Gene-Negative, TPS ≥10% Locally Advanced or Metastatic Non-Small Cell Lung Cancer
Brief Title: A Study to Evaluate the Safety and Tolerability of SCTB14 as First-Line Therapy in Non-Small Cell Lung Cancer.
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sinocelltech Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SCTB14-A301
Record Dates: First submitted 2026-01-09; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Non-Small Cell Lung Carcinoma (NSCLC)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — pembrolizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SCTB14 (Experimental): intravenous infusion on Day 1 of each 3-week cycle
  Interventions: Drug: SCTB14
- Pembrolizumab (Active Comparator): 200mg, intravenous infusion on Day 1 of each 3-week cycle
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: SCTB14 — SCTB14 is administered at selected dose by intravenous infusion on Day 1 of each 3-week cycle.
  Arms: SCTB14
Drug: Pembrolizumab — Pembrolizumab is administered at a fixed dose of 200 mg by intravenous infusion on Day 1 of each 3-week cycle.
  Arms: Pembrolizumab

SUMMARY:
This Phase III, randomized, double-blind study compares the efficacy and safety of SCTB14 versus pembrolizumab as first-line treatment in patients with driver gene-negative, TPS ≥10% locally advanced or metastatic non-small cell lung cancer (NSCLC). The primary objective is to assess superiority of SCTB14 over pembrolizumab in prolonging progression-free survival. Safety will be closely monitored.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign the written informed consent form prior to screening.
2. Age ≥ 18 years, both male and female.
3. ECOG Performance Status score of 0 to 1.
4. An expected survival of ≥ 3 months.
5. Histologically or cytologically confirmed, unresectable locally advanced (Stage IIIB/IIIC) or metastatic (Stage IV) Non-Small Cell Lung Cancer (NSCLC) that is not amenable to curative surgery or radical concurrent/sequential chemoradiotherapy.
6. For subjects with non-squamous cell carcinoma, as well as non-smoking subjects with squamous cell carcinoma containing mixed adenocarcinoma components, confirmation of the absence of EGFR sensitizing mutations or ALK gene rearrangements from tumor tissue is required prior to enrollment.
7. Subjects must provide a histology sample suitable for PD-L1 testing, with a Tumor Proportion Score (TPS) ≥ 10%.
8. No prior systemic anti-tumor therapy for the studied disease.
9. At least one measurable non-CNS lesion according to RECIST v1.1 criteria.
10. Adequate function of major organs.

Exclusion Criteria:

1. Known actionable driver gene mutations such as ROS1 fusion, BRAF V600E mutation, NTRK fusion, MET exon 14 skipping mutation, and RET fusion mutation.
2. Received non-specific immunomodulatory therapy or immunosuppressive drugs within 2 weeks before the first dose; received traditional Chinese medicine with antineoplastic indications within 1 week before the first dose.
3. Prior thoracic radiotherapy; or local anti-tumor therapy within 2 weeks before first dosing.
4. Prior treatment with antitumor immunotherapy, antiangiogenic therapy, or other small molecule tyrosine kinase inhibitor (TKI)-based antitumor drugs.
5. subjects with metastasis or compression involving the brainstem, meninges, or spinal cord, or those with active CNS metastases or multiple brain metastases.
6. Imaging demonstrates tumor invasion of major blood vessels, significant necrosis or cavitation within the primary tumor lesions, or the presence of lymphangitic carcinomatosis.
7. Imaging demonstrates tumor invasion or compression of adjacent vital organs or carries a risk of developing an esophagotracheal fistula or esophagopleural fistula.
8. History of hypertensive crisis or hypertensive encephalopathy, or the presence of uncontrolled hypertension despite medication, or poorly controlled diabetes despite pharmacotherapy.
9. A history of arterial thrombosis, deep vein thrombosis, cerebral infarction, transient ischemic attack, or significant vascular disease within 6 months prior to enrollment.
10. A history of myocardial infarction, unstable angina, cardiac insufficiency with New York Heart Association (NYHA) class ≥ III, or severe arrhythmia uncontrolled by medication within 6 months prior to enrollment.
11. The presence of any active autoimmune disease or a history of autoimmune disease with an anticipated recurrence.
12. A history of esophageal/gastric varices, severe ulcer, abdominal fistula, intra-abdominal abscess, gastrointestinal perforation and/or fistula, acute gastrointestinal bleeding, intestinal obstruction, or extensive intestinal resection within 6 months prior to the first dose.
13. A history of bleeding tendency, high bleeding risk, or coagulation dysfunction,.
14. The presence of other malignant tumors.
15. Toxicities from prior neoadjuvant/adjuvant therapy, surgery, radiotherapy, or other previous antitumor treatments have not recovered to Grade 0-1.
16. Receipt of a live or attenuated vaccine within 4 weeks prior to the first dose, or a plan to receive a live or attenuated vaccine during the study period; however, the use of inactivated vaccines is permitted.
17. Presence of any of the following infectious conditions: a) severe infection within 4 weeks prior to the first dose; b) active infection within 2 weeks prior to enrollment; c) active tuberculosis; d) positive HIV antibody; e) active hepatitis B or C; f) known active syphilis.
18. Major surgery planned or anticipated during the study period, or unhealed tissue present before enrollment..
19. Presence of symptomatic or recurrent pleural effusion, pericardial effusion, or ascites requiring drainage.
20. A history of non-infectious pneumonia requiring treatment or the presence of interstitial lung disease
21. A history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation.
22. Known hypersensitivity to any component of the investigational drug or a documented history of severe hypersensitivity reactions to any other monoclonal antibody.
23. Current participation in another clinical trial, with the exception of observational (non-interventional) studies or the follow-up phase of an interventional trial.
24. Pregnancy or lactation in female subjects.
25. A known history of alcohol or drug addiction, psychiatric disorders, or drug abuse in the subject.
26. Tumor-induced conditions or symptoms associated with a high medical risk.
27. Any other condition deemed by the investigator to be inappropriate for enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 246 (Estimated)
Dates: Start 2025-12-30 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) Assessed by Blinded Independent Central Review | Up to approximately 1.5 years
  Time from randomization to first documented progression or death (whichever occurs first).

SECONDARY OUTCOMES:
overall survival | Up to approximately 5 years
  The time from the date of randomization to the date of death from any cause.
Progression-Free Survival (PFS) as Assessed by Investigator | Up to approximately 1.5 years
  Time from randomization to first documented progression or death (whichever occurs first).
Confirmed Objective Response Rate (ORR) Assessed by Blinded Independent Central Review | Up to approximately 1.5 years
  The proportion of subjects with a best overall confirmed response of Complete Response (CR) or Partial Response (PR)
Disease Control Rate (DCR) Assessed by Blinded Independent Central Review | Up to approximately 1.5 years
  The proportion of patients with a best overall response of Complete Response (CR), Partial Response (PR), or Stable Disease (SD).
Duration of Response （DOR）Assessed by Blinded Independent Central Review | Up to approximately 1.5 years
  The time from the first documented objective response (Complete Response [CR] or Partial Response [PR]) to the first documented disease progression or death from any cause, whichever occurs first.
Time to Response (TTR) | Up to approximately 1.5 years
  Time from the date of randomization to the first documented objective response (Complete Response [CR] or Partial Response [PR]
Treatment-Emergent Adverse Event（TEAE） | The first dose of study drug until 30 days (±7 days) after the last dose
  Any adverse event that occurs or worsens in severity after the initiation of study drug administration
Serious adverse events (SAEs) | From the first dose of study druguntil 60 days after the last dose.
  An adverse medical event occurring after a subject receives the investigational drug that results in any of the following outcomes: death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, or is a congenital anomaly/birth defect.
immune-related adverse events (irAEs) | From the first dose of study druguntil 60 days after the last dose
  All grades of adverse drug reactions (ADRs) that occur after a subject receives the investigational drug and are assessed as having a causal relationship to an immune-mediated mechanism.
PD-L1 expression | Up to approximately 1.5 years.
  The correlationship between PD-L1 expression and anti-tumor activity.
Quality of Life Questionnaire | Up to approximately 1.5 years.
  Change in Health-Related Quality of Life EORTC QLQ-C30
Quality of Life Questionnaire | Up to approximately 1.5 years
  Change in Health-Related Quality of Life QLQ-LC13
Anti-drug antibodies (ADA) | Up to approximately 1.5 years
  Number and percentage of subjects with anti-drug antibodies (ADA) to SCTB14
Pharmacokinetic (PK) | Up to approximately 1.5 years.
  Serum concentration of SCTB14 at different time points

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Chest Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No